CLINICAL TRIAL: NCT00201591
Title: Which Training Intensity is Most Effective in Improving Myocardial Function in Patients With Coronary Artery Disease?
Brief Title: Training at Different Intensities in Coronary Artery Disease -Effects on Myocardial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trehab I NTNU
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Exercise training; Intensity; Randomized; echocardiography; Aerobic Exercise
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Exercise training for 10 weeks

SUMMARY:
The study investigated if aerobic endurance exercise of different intensity has different impact on the physical capacity and myocardial function in patients with coronary artery disease. Patients with stable CAD trained for 10 weeks, and oxygen consumption and myocardial function were measured before and after this period. Patients were randomly assigned to each exercise group.

DETAILED DESCRIPTION:
Peak oxygen consumption was measured by gas-analysis. Myocardial function was measured by echocardiography. Exercise was performed on treadmills under close supervision of an exercise physiologist. Patients had to complete over 70% of sessions to be included in analysis. Three sessions were scheduled every week. Heart rate (HR) was about 85 % of max HR in the high intensity group, and about 65 % in the moderate intensity group.

ELIGIBILITY:
Inclusion Criteria:

* stable coronary artery disease
* over 4 months since cardiovascular event

Exclusion Criteria:

* heart failure
* inability to exercise

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2002-08; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption

SECONDARY OUTCOMES:
Quality of life
Myocardial function measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Stig A Slørdahl, Prof, Study Chair — Norwegian University of Science and Technology
Locations (1):
- Dept. of Circulation and Medical Imaging, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Amundsen BH, Rognmo O, Hatlen-Rebhan G, Slordahl SA. High-intensity aerobic exercise improves diastolic function in coronary artery disease. Scand Cardiovasc J. 2008 Apr;42(2):110-7. doi: 10.1080/14017430701744477. PMID 18365893